CLINICAL TRIAL: NCT03844555
Title: Open Label, Phase I Study to Assess and Compare the Pharmacokinetic Parameters After Single Oral Administration of Elafibranor 120 mg in Renal Impaired Patients and Healthy Subjects With Normal Renal Function
Brief Title: Elafibranor Pharmacokinetic Parameters in Renal Impaired Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genfit (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GFT505-118-13; 2018-002481-39 (EudraCT Number)
Record Dates: First submitted 2019-02-15; First posted 2019-02-18 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Renal Impairment; Renal Insufficiency; Kidney Diseases; Pharmacokinetics
MeSH Terms: conditions — Renal Insufficiency; Kidney Diseases | interventions — 2-(2,6-dimethyl-4-(3-(4-(methylthio)phenyl)-3-oxo-1-propenyl)phenoxyl)-2-methylpropanoic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- End Stage Renal Disease (Experimental): Single oral dose of elafibranor 120mg
  Interventions: Drug: Elafibranor
- Healthy (Experimental): Single oral dose of elafibranor 120mg
  Interventions: Drug: Elafibranor

INTERVENTIONS:
Drug: Elafibranor — 120mg oral single dose
  Other Names: GFT505

SUMMARY:
This study is being conducted in order to assess the need for dose adjustment for elafibranor in participants with renal impairment. Pharmacokinetic parameters of elafibranor and its active metabolite (GFT1007) will be compared in severe renal impaired participants (eGFR<15mL/mn/1.73m^2) versus healthy participants after a single oral administration of elafibranor 120 mg

ELIGIBILITY:
Inclusion Criteria:

For all participants

1. Male or female subjects, aged 18 to 75 years inclusive;
2. Females participating in this study must be of non-childbearing potential or using highly efficient contraception for the full duration of the study
3. Negative serum pregnancy test at screening (if applicable);
4. Non-smoker subject or smoker of not more than 5 cigarettes a day;

   For Renally Impaired Participants
5. ESRD patient not yet on dialysis with an estimated glomerular filtration rate (eGFR) <15mL/min/1.73m^2;
6. Documented renal impairment indicated by reduced eGFR within 12 months of screening or longer;
7. Stable renal function as evidenced by ≤ 30 percent difference in two evaluation of eGFR on two separate occasions separated by at least 28 days with one measurement being the value at screening;
8. Body Mass Index (BMI) between 20 and 36 kg/m^2 inclusive.

   For Healthy Volunteers with normal renal function:
9. eGFR ≥ 90mL/min/1.73m^2;
10. No proteinuria (< 0.15 g/L determined by urinalysis);
11. Body Mass Index between 20 and 30 kg/m^2 inclusive and body weight not lower than 55kg;
12. Matched to at least 1 renal impaired patient by ethnic group, sex, age (+/- 10 years) and BMI (+/- 20 percent).

Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

All Participants

1. Positive Hepatitis B surface antigen or anti Hepatitis C Virus antibody, or positive results for Human Immunodeficiency Virus 1 or 2 tests;
2. History or presence of drug or alcohol abuse (alcohol consumption > 40 grams/day);
3. Blood donation (including in the frame of a clinical trial) within 2 months before administration or blood donation planned during the study or within 2 months following participation to the study;
4. Participants who are pregnant or breastfeeding. Participants should not be enrolled if they plan to become pregnant during the time of study participation;
5. Positive results of screening for drugs of abuse;
6. Evidence or history of clinically significant uncontrolled hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, metabolic, systemic, infectious, or allergic disease (including drug hypersensitivity or allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing);
7. General anesthesia within 3 months before administration;
8. Major surgery within 28 days prior to randomization or major surgery planned during the next 6 months.

   For Renally Impaired Participants:
9. History of renal transplant;
10. Evidence of an unstable clinically important medical condition other than impaired renal function;
11. Acute exacerbation or unstable renal function, as indicated by worsening of clinical and/or laboratory signs of renal impairment, within the 4 weeks before study drug administration;
12. Participants undergoing any method of dialysis or hemofiltration;
13. Disorders or surgery of the gastrointestinal tract which may interfere with drug absorption or may otherwise influence the pharmacokinetics of the investigational medicinal product (e.g., inflammatory bowel disease, resections of the small or large intestine, etc.);
14. History of febrile illness within 5 days prior to dosing;
15. Evidence of clinically significant liver disease or liver damage (e.g., hepatitis B or C, autoimmune hepatitis, primary biliary cirrhosis, non-alcoholic fatty liver disease, elevated aspartate aminotransferase or alanine aminotransferase that is considered clinically significant by the Investigator, etc.). Presence or history of protein drug hypersensitivity, or allergic disease diagnosed and treated by a physician
16. Any drug intake during the 2 weeks or 5 half-life of the drug preceding the first administration except those defined in the protocol

    For Healthy Volunteers with normal renal function:
17. Any history or presence of renal disease
18. Frequent headaches (> twice a month) and / or migraines, recurrent nausea and / or vomiting;
19. Symptomatic hypotension whatever the decrease of blood pressure or asymptomatic postural hypotension defined by a decrease in Systolic Blood Pressure (≥20 mmHg) or Diastolic Blood Pressure (≥10 mmHg) within three minutes when changing from the supine to the standing position;
20. Inability to abstain from intensive muscular effort;
21. Any drug intake (except paracetamol 3g/d or contraception) during the 2 weeks or 5 half-life of the drug preceding the first administration;
22. Subject who would receive more than 4500 euros as indemnities for his participation in biomedical research within the 12 last months, including the indemnities for the present study.

Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-21 (Actual)

PRIMARY OUTCOMES:
Area under curve from dosing time to last measurement (AUC(0-t)) of elafibranor and active metabolite | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose
  In participants with end stage renal disease compared to healthy volunteers
Area under curve from dosing time to infinity (AUC(0-∞)) of elafibranor and active metabolite | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose
  In participants with end stage renal disease compared to healthy volunteers

SECONDARY OUTCOMES:
Plasma pharmacokinetics: maximum plasma drug concentration (Cmax) | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose
  for elafibranor and metabolites
Plasma pharmacokinetics: elimination half-life (t1/2) | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose
  for elafibranor and metabolites
Plasma pharmacokinetics: apparent volume of distribution (Vd/F) | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose
  for elafibranor
Plasma pharmacokinetics: renal clearance (CLr) | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose
  for elafibranor and metabolites
Plasma pharmacokinetics: apparent non renal clearance (CLnr/F) | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose
  for elafibranor
Plasma pharmacokinetics: apparent total clearance (CL/F) | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose
  for elafibranor
Plasma pharmacokinetics: area under the plasma concentration-time curve extrapolated from time t to infinity as a percentage of total area under the plasma concentration-time curve (%AUCextra) | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose
  for elafibranor and metabolites
Plasma pharmacokinetics: area under curve from dosing time to last measurement (AUC(0-t)) of glucuronide metabolites and corresponding aglycones | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose
  for the glucuronide metabolites of elafibranor and corresponding aglycones
Plasma pharmacokinetics: area under curve from dosing time to infinity (AUC(0-∞)) of glucuronide metabolites and corresponding aglycones | pre-dose and at 0.17, 0.33, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 and 216 hours post-dose
  for the glucuronide metabolites of elafibranor and corresponding aglycones
Urine pharmacokinetics: amount excreted (Ae) | pre-dose and then 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  for elafibranor and metabolites, if applicable. 24 hours urine collection from dosing to 216 hours post-dose
Urine pharmacokinetics: cumulative amount excreted (Ae0-t) | pre-dose and then 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  for elafibranor and metabolites, if applicable. 24 hours urine collection from dosing to 216 hours post-dose
Urine pharmacokinetics: percentage of dose excreted (Fe) | pre-dose and then 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  for elafibranor and metabolites, if applicable. 24 hours urine collection from dosing to 216 hours post-dose
Urine pharmacokinetics: cumulative percent of dose excreted (Fe0-t) | pre-dose and then 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  for elafibranor and metabolites, if applicable. 24 hours urine collection from dosing to 216 hours post-dose
Urine pharmacokinetics: renal clearance (CLR) | pre-dose and then 24, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  for elafibranor and metabolites, if applicable. 24 hours urine collection from dosing to 216 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Birman, MD, Study Director — Genfit
Locations (2):
- Eurofins Optimed, Gières, France
- ARENSIA Exploratory Medicine Unit, Nephrology Hospital Dr. Carol Davilla, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No